CLINICAL TRIAL: NCT00965939
Title: Study to Assess Response to Tamoxifen in (cT3)/ Inoperable Locally Advanced / Metastatic ER-positive Breast Cancer by the 'Tamoxifen Activity Score' Based on Drug Interaction and Polymorphisms in Genes Coding for Tam. Metabolising Enzymes.
Brief Title: An Observational Study to Assess Response to Tamoxifen in Breast Cancer Patients
Acronym: CYPTAMBRUT-2
Status: Completed | Type: Observational
Sponsor: Vlaamse Vereniging voor Obstetrie en Gynaecologie (Other)
Responsible Party: Sponsor
Other Study IDs: S51257; B32220095818
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: ER-positive Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
CYPTAM-BRUT 2 is a prospective, multicentric study including postmenopausal women receiving tamoxifen for metastatic, locally advanced (stage IIIB/C) or in the neoadjuvant setting for measurable estrogen-receptor positive breast cancers. The primary endpoint is the difference in efficacy of tamoxifen, defined as the objective response rate using RECIST criteria, between women with a normal versus low Tamoxifen Activity Score (TAS) after 3-6 months of tamoxifen use. The TAS score is based on the presence of genetic variations and drug interactions. Secondary endpoints are time to progression, clinical benefit, serum metabolite concentrations, endometrial changes and menopausal symptoms. Patients using tamoxifen in the neoadjuvant setting needs being operated between 4-6 months following the start of tamoxifen.

DETAILED DESCRIPTION:
This multi-centre open label single arm non randomized observational study will compare the efficacy in terms of overall response rate and progression free survival of tamoxifen as first line therapy in 3 groups of postmenopausal women with measurable hormone dependent large, locally advanced or metastatic breast cancer. The 3 groups are women with a normal and those with a low 'tamoxifen activity score' based on genetic polymorphisms for CYP2D6 and other genes that are important in the metabolism of tamoxifen using SEQUENOM's MassARRAY technology.

The study is subject to Ethical Commission approval and patient consent. The study will necessitate collection of blood for genetic analyses.

We will investigate the relation between the studied genotype, the use of drugs that interfere with tamoxifen and tamoxifen-related endpoints like regression of metastatic or locally advanced or large oestrogen receptor positive breast cancer in tamoxifen users. The 'tamoxifen activity score' has been used by a group in the US showing a link with tamoxifen compliance. The score will be adapted to the Belgian situation based on the prevalence of polymorphism in a Belgian population. The efficacy of tamoxifen will be correlated with a predefined 'tamoxifen activity score' which is based on the presence of single nucleotide polymorphisms (SNP) in relevant genes combined with the effect of well known drugs that interfere with the metabolism of tamoxifen.

The study will be conducted in several clinical sites in Belgium. All patients will receive tamoxifen 20mg daily. Patients with a large operable or inoperable non-metastatic breast cancer will be considered for surgery no more than 4 months on tamoxifen. If operable, they will postoperatively receive the most appropriate adjuvant therapy and for hormone therapy either continue tamoxifen or receive an oral aromatase inhibitor as decided by the clinician. If women with a locally advanced inoperable breast cancer are not operable after the 4 months of neo-adjuvant therapy, another appropriate salvage therapy will be proposed. Women with metastatic breast cancer will continue treatment until clinical or imaging progression or unacceptable toxicity development. Patients that experience progression of their disease as defined by RECIST criteria will receive salvage therapy by an oral aromatase inhibitor if tamoxifen is given in first line but some patients may require another therapy like chemotherapy. The study will require approximately 14 months to recruit and another 7 months to events/data analyses as the estimated time to progression in this setting is 9-12 months if tamoxifen is given as first line endocrine therapy for those in the metastatic setting

ELIGIBILITY:
Inclusion Criteria:

* - Female > 18 years of age
* Written and voluntary informed consent understood signed and dated
* Histologically or cytologically confirmed measurable invasive adenocarcinoma of the breast either large (cT3), locally advanced stage IIIB/C inoperable, or metastatic and not amenable to curative therapy with surgery or radiotherapy.
* Measurable disease is defined as follows: CT scan for metastatic or locally advanced stage IIIB disease and ultrasound of the breast for operable large size breast cancers where tamoxifen is given for neoadjuvant endocrine therapy .
* Patients must be postmenopausal as defined by criteria in appendix 1.
* Breast cancer should be considered as oestrogen receptor positive by the clinician using immunohistochemistry readings as is standard procedure for local pathologist
* Prior endocrine tamoxifen therapy in the adjuvant setting is allowed if there is more than 12 months after completion of adjuvant tamoxifen.
* Prior radiotherapy is allowed but evaluable lesions that have been irradiated need to be progressive before starting in the study
* Concurrent use of bisphosphonates is allowed if they are started 2 weeks before study start and these drugs should be continued as planned throughout the study
* Adequate renal and liver function Serum creatinine and serum bilirubin ≤ 1.5 X ULN Serum ALT and AST ≤ 2.5 X ULN (or ≤ 5 in case of liver metastases)
* Serum calcium should be ≤ 11,6 mg/dl
* ECOG performance status 0,1,2 (appendix 2)

Exclusion Criteria:

* - Male
* Life threatening disease requiring a quick response (eg, extensive hepatic or pulmonary involvement)
* CNS involvement
* Less than 12 months since stopping tamoxifen in the adjuvant setting
* Previous chemotherapy, tamoxifen or more than one line hormone therapy or targeted therapy for locally advanced/ metastatic breast cancer
* Bone lesions only
* One line of prior endocrine therapy with an oral aromatase inhibitor for locally advanced or metastatic breast cancer is not allowed also not if there is clear progression according to RECIST and the clinician judges tamoxifen an appropriate second line therapy
* Contra indication for tamoxifen: history of DVT/vaginal bleeding of unknown origin
* Dementia
* History of other malignancy that may interfere with at least 6 months of tamoxifen therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female, with ER-positive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-02; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
ORR | 3 months/ 6 months

SECONDARY OUTCOMES:
TTP | 3 months/ 6 months
clinical benefit (CR + PR + SD ≥ 6 months) | 3 months/6months
Endometrial thickness and uterine volume | Baseline/ 3 months
Tolerability of tamoxifen-HRQoL questionnaire | baseline/ 3months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Neven, Principal Investigator — UZ Leuven
Locations (12):
- Belgium (12):
  - Imelda ziekenhuis, Bonheiden, Antwerpen
  - AZ St-Maarten Campus Rooienberg, Duffel, Antwerpen
  - Heilig-Hartziekenhuis, Lier, Antwerpen
  - Ziekenhuizen Oost-Limburg campus St-jan, Genk, Limburg
  - Virga Jesse Ziekenhuis, Hasselt, Limburg
  - AZ St-Blasius, Dendermonde, Oost-Vlaanderen
  - Maria-Middelares, Ghent, Oost-Vlaanderen
  - UZ, Ghent, Oost-Vlaanderen
  - AZ St-Nikolaas, St-Niklaas, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - Heilig-Hartziekenhuis, Roeselare, West-Vlaanderen
  - UCL, Brussels